CLINICAL TRIAL: NCT00693017
Title: A Double-blind, Randomised, Placebo-controlled, Multi-centre Study to Assess the Efficacy and Safety of Adjunctive Zonisamide in Myoclonic Seizures Associated With Idiopathic Generalised Epilepsy
Brief Title: Efficacy and Safety of Adjunctive Zonisamide in Myoclonic Seizures Associated With Idiopathic Generalised Epilepsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2090-E044-317; 2007-003556-10 (EudraCT Number)
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Zonisamide (Active Comparator)
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — 50-400 mg capsules once daily in the evening orally.
  Maximum study duration 28 weeks comprising:
  Baseline Period (Week -8 to Week 0): no treatment
  Titration Period (Week 0 to Week 4): 50 mg daily titrated weekly until 300 mg was reached by Week 4
  Maintenance Period (Week 4 to Week 16) 400 mg (or 350 mg in the event of dose limiting adverse events)
  Down Titration Period (4 Weeks)
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Placebo — 50-400 mg Zonisamide Placebo capsules once daily in the evening orally.
  Maximum study duration 28 weeks comprising:
  Baseline Period (Week -8 to Week 0): no treatment
  Titration Period (Week 0 to Week 4): 50 mg Zonisamide Placebo daily titrated weekly until 300 mg was reached by Week 4
  Maintenance Period (Week 4 to Week 16) 400 mg Zonisamide Placebo (or 350 mg in the event of dose limiting adverse events)
  Down Titration Period (4 Weeks)
  Arms: Placebo

SUMMARY:
This study is intended to provide evidence that zonisamide is safe and effective in the treatment of myoclonic seizures. The total planned trial duration will be 6.5 months. After that, subjects who have completed the study will be eligible to enroll in an open-label extension study until zonisamide is marketed for this indication or further development in this indication stops. This extension study will be described in a separate protocol (E2090-E044-318).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and aged 12-65 years.
2. Subject has at least eight days with at least one myoclonic seizure over the two months Baseline Period. Myoclonic seizures must occur in the context of IGE and may be accompanied by other primary generalized seizures, provided these are also consistent with a diagnosis of Idiopathic Generalized Epilepsy (IGE).
3. Subject (or parent/caregiver, for subjects below the age of consent) is willing to sign an informed consent form. Subjects below the age of consent in their country, must where appropriate be willing to give informed (written or verbal) assent. Subjects from the age specified in local regulations will be required to sign an appropriate informed consent form.
4. Subject is taking a stable regimen of one or two other AEDs for at least two weeks prior to Visit 1 (start of the Baseline Period).
5. Subject has a clinical diagnosis of any type of idiopathic generalised epilepsy (IGE) which has myoclonic seizures (and which may be accompanied by other generalised seizure types), according to the International League Against Epilepsy (ILAE) Classification of Epileptic Seizures (1981) and the ILAE Classification of Epilepsies and Epileptic Syndromes (1989). Diagnosis should have been established by clinical history, electroencephalogram (EEG) and computed tomography/magnetic resonance imaging (CT/MRI) of the brain consistent with idiopathic generalised epilepsy. A CT/MRI scan should have been performed within five years of the screening visit or, if not available from this period, should be performed in the Baseline Period.
6. EEG should have been performed within one year of the screening visit or, if not available from this period, should be performed in the Baseline Period.
7. Female subjects are pre-menarchal, or if of childbearing potential, are not pregnant or lactating, or are post-menopausal.
8. Female subjects of childbearing potential ≥ 18 years must abide by one of the following medically acceptable contraceptive measures: oral contraception pill, contraceptive injections, implants or patches, intrauterine device in place for at least three months or vasectomised partner or abstinence throughout the study. Subjects <18 years and of childbearing potential must be either abstinent or willing to use one of the medically appropriate forms of contraception for the duration of the study.

Exclusion Criteria:

1. Subject has progressive or focal neurological disease (as determined by preexisting brain imaging such as CT or MRI performed maximally five years before the screening visit), or clinically significant organic disease.
2. Subject has a history of, or results of clinical investigations (including EEG data) that are suggestive of, partial seizures as defined by the ILAE, including generalised tonic clonic seizures which are suspected to be secondarily generalised.
3. Subjects with cryptogenic or symptomatic generalised epilepsy.
4. Subjects with psychogenic seizures.
5. Subject has a history of convulsive status epilepticus within a year of screening while complying with AEDs.
6. Subject has a history of renal calculi or renal insufficiency (above the upper normal limits of creatinine).
7. Subject has a known diagnosis of human immunodeficiency virus (HIV) or hepatitis B or C.
8. Subject has a predisposing condition that might interfere with absorption, distribution, or excretion of zonisamide.
9. Subject has a history of sensitivity to sulfonamide drugs or to zonisamide or any of its excipients.
10. Subject has a recent history of excessive alcohol use or drug abuse.
11. Subject has a history of suicide attempt in the five years before the screening visit.
12. Subject has abnormal screening laboratory values that are clinically significant.
13. Subject has a history of demonstrated non-compliance with treatment, or the subject or parent/caregiver can be reasonably expected not to be compliant with study procedures or to complete the study.
14. Subject has participated in a study of an investigational drug or device within 30 days prior to screening.
15. Subject has received previous treatment with zonisamide.
16. Subject is treated with ketogenic diet or vagus nerve stimulator.
17. Subject has a history of necessary treatment with rescue benzodiazepines which is foreseen to continue during the study. Rescue benzodiazepines will not be allowed in this study (stable dosing with a benzodiazepine as (one of the) baseline anti-epileptic drug(s) is allowed).
18. Concomitant use of acetazolamide, carbonic anhydrase inhibitors such as topiramate and drugs with anticholinergic activity.
19. Current psychosis or moderate to severe depression, or use of anti-psychotic drugs, MAOIs, tricyclic antidepressants, benzodiazepine or barbiturate treatment for disorders other than epilepsy, and stimulants (amphetamine derivatives) within 28 days before the screening visit.
20. Concomitant use of felbamate or use of felbamate within two months prior to Visit 1.
21. Subject is unable to swallow capsules.
22. Subject is not in general good health as determined by medical history, physical exam and screening laboratory results.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob van Maanen, M.D., Study Director — Eisai Limited
Locations (71):
- Australia (4):
  - Strategic Health Evaluators Pty Ltd, Chatswood, New South Wales
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Austin Health, Heidelburg, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
- Croatia (3):
  - CH Split, Split, HR
  - CH Sestre Milosrdnice University Hospita, Zagreb, HR
  - UHC Zagreb, Zagreb, HR
- Czechia (7):
  - Neurologicke oddeleni, Kralove
  - Private Neurologi Office, Kroměříž
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice s poliklinikou Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Pilsen
  - Nemocnice Na Homolce, Prague
  - Centrum neurologicke pece, Rychnov nad Kněžnou
- Estonia (3):
  - West-Tallinn Central Hospital, Tallinn
  - Neurodiagnostica AP OY, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Kuopio Epilepsy Center, Kuopio
  - Oulu University Central Hospital, Oulu
- Germany (5):
  - Institut fur Diagnostik der Epilepsien (IDE) gGmbH Epilepsie-Zentrum Berlin- Brandenburg., Berlin
  - Neurochirurgische Klinik der Universitat Freiburg, Freiburg im Breisgau
  - Interdisziplinares Epilepsiezentrum am Klinikum der Philipps-Universitat Marburg, Marburg
  - Neurologische Gemeinschaftspraxis, München
  - Universitatsklinikum Ulm, Ulm
- Hungary (9):
  - National Institute of Psychiatry and Neurology, Budapest
  - Heim Pal Hospital, Budapest
  - Szent Istvan Hospital, Budapest
  - Orszagos Idegsebeszeti Tudomanyos Intezet, Budapest
  - Bethesda Hospital for Children, Budapest
  - Bekes County Pandy Kalman Hospital, Gyula
  - Bacs-Kiskun County ONK Hospital, Kecskemét
  - Vas County Markusovszky Hospital, Szombathely
  - Veszprem County Csolnoky F. Hospital, Veszprém
- Lithuania (3):
  - Kaunas Medical University Hospital, Kaunas
  - Neuromeda, Kaunas
  - Vilnius University Hospital Santariskiu klinikos, Vilnius
- Poland (6):
  - Niepubliczny ZOZ Kendron, Bialystok
  - Wojewozki Szpital Specjalistyczny im. M. Kopernika, Gdansk
  - Specjalistyczny Szpital Wieloprofilowy, Katowice
  - Centrum Neurologii Klinicznej, Krakow
  - Szpital im. M. Kopernika, Lodz
  - Uniwersytet Medyczny, Poznan
- Romania (7):
  - Centrul Medical Sana, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta "Sf Spiridon" Iasi, Lasi
  - Spitalul Clinic de Urgenta "Sfanta Treime", Lasi
  - Spitalul Clinic Judetean de Urgenta Tg Mures, Tg Mures
- Russia (11):
  - GOU VPO Krasnoyarskaya State Medical Academy of Roszdrav, Krasnoyarsk
  - FGU Moscow Research Institute of Psychiatry of Roszdrav, Moscow
  - GOU VPO Russian State Medical University of Roszdrav, Moscow
  - GUZ of Moscow City Clinical Hospital #1 n.a. N.I.Pirogov, Moscow
  - GOU VPO Moscow State University of Medicine and Dentistry of Roszdra, Moscow
  - GOU VPO Novosibirsk State Medical University of Roszdrav, Novosibirsk
  - GU St. Petersburg Research Institute of Psychoneurology Bekhtereva of Roszdrav, Saint Petersburg
  - St. Petersburg State Medical Pediatric Academy, Saint Petersburg
  - GOU VPO St. Petersburg State Medical University, Saint Petersburg
  - GOU VPO Smolensk State Medical Academy of Roszdrav, Smolensk
  - Yaroslavskaya State Medical Academy, Yaroslavl
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - University Medical Center Zvezdara, Belgrade
  - Clinical center Kragujevac, Kragujevac
  - Clinical Center of NIS, Niš
- Ukraine (7):
  - Tsentr Psihosomatychnoyi Patologiyi Dnipropetrovskoyi oblasnoyi klinichnoyi likarni imeni Mechnikova, Dnipropetrovsk
  - Derzhavna Ustanova Institut Nevrologiy, Kharkiv
  - Kyiv City Psychiatric Hospital #2, Poliklinichne Viddilenya, Kyiv
  - Miska Klinichna psihonevrologichna, Kyiv
  - Lvivskyiy oblasnyi Protyepileptuchnyy tsentr, Lviv
  - Odesskyy Derzhavnyy Medychnyy Universitet, Odesa
  - Vinnitskyy Natsionalnyy Medychnyy Universitet, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at three study centers (1 in Australia and 2 in Hungary). A further 39 study centers in Europe and Australia were initiated. A total of 12 study sites in the following countries were not initiated; (2 in Finland), (3 in Czech Republic), and (7 in Ukraine) during the period of 04 June 2008 to 05 January 2009.
Pre-assignment Details: 10 participants were screened for eligibility and six participants did not continue after the Screening Visit due to the Sponsor's decision to terminate the study. 4 participants were enrolled and treated during the study.
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Sponsor Decision | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (16.97) | 33.5 (23.33) | 28.8 (17.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Considered Responders as Assessed During the Maintenance Period
Description: The number of participants who were considered responders during the 12 week Maintenance Period (Week 4 to Week 16). A responder was defined as a participant with a decrease >= 50% from baseline in the number of days with myoclonic seizures per 28 days (i.e. 28-day myoclonic seizure frequency in Period from Week 4 to the Week 16 visit compared to Week -8 to randomization at Week 0 [Screening/ Baseline Period]). Occurrence of seizures was documented in a seizure diary. The diary was dispensed at the Screening Visit and maintained by the participant (parent/caregiver) and reviewed at each following visit. The diary was completed daily. All seizures except myoclonic seizures were counted individually in the the diary. Due to early termination of the study by the Sponsor, no formal analyses were conducted.
Time Frame: Baseline (Week -8 to Week 0) and Maintenance Period (Week 4 to Week 16)
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage Change From Baseline in the Monthly Number of Days With Myoclonic Seizures
Description: Percentage Change from Baseline in the monthly number of days with myoclonic seizures was assessed both for the Maintenance Period alone (Week 4 to Week 16) and for the entire double-blind treatment period (Week 0 to Week 16). Due to early termination of the study by the Sponsor, no formal analyses were conducted.
Time Frame: Baseline and up to 16 weeks
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Zonisamide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=2) | Placebo (N=2)
Sudden unexplained death in epilepsy (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=2) | Placebo (N=2)
Vision blurred (Eye disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study by the Sponsor. No formal analyses were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No